CLINICAL TRIAL: NCT00985023
Title: A Randomized, Prospective Comparison of Stainless Steel and Bioabsorbable Screw Fixation of Lisfranc Foot Injuries
Brief Title: A Comparison of Stainless Steel and Bioabsorbable Screw Fixation of Lisfranc Foot Injuries
Acronym: Lisfranc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Principal Investigator, Jamal Ahmad, Assistant Professor of Orthopaedic Surgery, Rothman Institute Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lisfranc
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Unstable Lisfranc Fracture-dislocations of the Midfoot
Keywords: Unstable; Lisfranc; fracture; dislocation; midfoot
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steel screw fixation (Active Comparator)
  Interventions: Procedure: Steel screw fixation of Lisfranc fracture-dislocation.
- Bioabsorbable screw fixation (Experimental)
  Interventions: Procedure: Absorbable screw fixation of Lisfranc fracture-dislocations.

INTERVENTIONS:
Procedure: Steel screw fixation of Lisfranc fracture-dislocation. — Stainless steel screw fixation of unstable Lisfranc fracture-dislocations of the midfoot.
  Other Names: Steel screw
  Arms: Steel screw fixation
Procedure: Absorbable screw fixation of Lisfranc fracture-dislocations. — Bioabsorbable (poly-levo-lactic acid) screw fixation of unstable Lisfranc fracture-dislocations of the midfoot.
  Other Names: Smart Screw
  Arms: Bioabsorbable screw fixation

SUMMARY:
The Lisfranc ligaments are a group of ligaments that connect the bones of the middle portion of the foot to each other. The Lisfranc ligaments allow for a normal and stable range of motion and shape to the foot. In certain foot fractures where the Lisfranc ligaments are damaged, the constraint and stability it had given to the middle of the foot is lost. Attempted activity at the foot will result in pain and abnormal motion. If injury to the Lisfranc ligaments is left untreated, the eventual end result is foot arthritis and deformity.

The current standard orthopaedic treatment of foot fractures with Lisfranc ligament injuries is surgery. The foot fractures are fixed with metal screws. The Lisfranc ligaments are fixed by compressing the space between the middle bones of the foot with steel screws. These screws allow for ligament healing. As the ligaments heal, the patient should not resume activity with the fixed foot too soon as the screw may break. Upon breakage, the ligament repair may fail and the screw is now difficult to surgically remove. Regardless of breakage, a second surgical procedure is often recommended to remove the steel screw 6 months after foot surgery. This allows for a complete return of normal foot range of motion, but at the cost of a second surgical procedure.

The investigators hypothesize that absorbable screw fixation of the Lisfranc ligaments does not yield significant differences in postoperative foot stability, ligament function, and symptoms when compared to steel screw fixation. In addition, absorbable screw fixation of the Lisfranc ligaments offers the advantage that a second surgical procedure to remove the screw is not necessary.

DETAILED DESCRIPTION:
The Lisfranc ligaments are a group of ligaments that connect the bones of the middle portion of the foot to each other. The Lisfranc ligaments allow for a normal and stable range of motion and shape to the foot.

In certain foot fractures, the Lisfranc ligaments are damaged. When the Lisfranc ligaments are disrupted, the constraint and stability it had given to the middle of the foot is lost. Attempted activity at the foot will result in pain and abnormal motion. If injury to the Lisfranc ligaments is left untreated, the eventual end result is foot arthritis and deformity.

The current standard orthopaedic treatment of foot fractures with Lisfranc ligament injuries is surgery. The foot fractures are fixed with metal screws. The Lisfranc ligaments are fixed by compressing the space between the middle bones of the foot with steel screws. These screws allow for ligament healing. As the ligaments heal, the patient should not resume activity with the fixed foot too soon as the screw may break. Upon breakage, the ligament repair may fail and the screw is now difficult to surgically remove. Regardless of breakage, a second surgical procedure is often recommended to remove the steel screw 6 months after foot surgery. This allows for a complete return of normal foot range of motion, but at the cost of a second surgical procedure.

The use of materials that can be absorbed by the human body to fix the Lisfranc ligaments has only been studied in 1 paper. One such material is the Smart Screw (Bionx, Blue Bell, Pennsylvania) which is approved by the Food and Drug Administration (F.D.A.) and made of polylevolactic acid (PLA). Absorbable screws could be ideal for the treatment of Lisfranc ligament injuries. They can provide a mechanical scaffold to allow for ligament healing. They are absorbable which eliminates the need for a second surgery to remove a screw. They can be used for foot injuries where the rate of healing and thus absorption is rapid. Although, absorbable implants are weaker than metal implants, the absorbable screw can be protected from breaking by restricting weight bearing after surgery. If the absorbable screw does break, there is no need to remove the fragments in the foot bones as they are absorbable.

Comparing the long-term results of fixing the Lisfranc ligaments with either a steel or absorbable screw is important as there are no studies on the subject to date. There is only 1 published study regarding absorbable screws to fix the Lisfranc ligaments. The purpose of this study is to compare the outcome of steel and absorbable screw fixation of the Lisfranc ligaments in foot injuries in two surgeons' practice.

We hypothesize that absorbable screw fixation of the Lisfranc ligaments does not yield significant differences in postoperative foot stability, ligament function, and symptoms when compared to steel screw fixation. In addition, absorbable screw fixation of the Lisfranc ligaments offers the advantage that a second surgical procedure to remove the screw is not necessary.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be adults of any gender or race.
* The underlying diagnosis will be a Lisfranc foot injury.
* The indication for fixing the Lisfranc ligaments is abnormal separation of the middle part of the foot from each other.
* Subjects will have received either a steel or absorbable screw to fix the Lisfranc ligaments.

Exclusion Criteria:

* Subjects must not have intact or normal Lisfranc ligaments in the foot.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Return to pre-injury level of function. | 2 years

SECONDARY OUTCOMES:
Restoration of normal midfoot alignment and stability. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Ahmad, M.D., Principal Investigator — Rothman Institute Orthopaedics
Locations (2):
- United States (2):
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Nazareth Hospital, Philadelphia, Pennsylvania